CLINICAL TRIAL: NCT02198586
Title: Apoe Impact Study on Brain Structure and Function, in a Population 45 to 75 Years Old
Status: Completed | Type: Observational
Sponsor: Barcelonabeta Brain Research Center, Pasqual Maragall Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: MRI/FBB 2014
Record Dates: First submitted 2014-07-15; First posted 2014-07-23 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's, MRI, APOE
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No treatment: The population of this study is 45 to 75 years old at the time of inclusion in the parent study (ClinicalTrials.gov ID: NCT01835717).

SUMMARY:
The purpose of this study is to investigate the influence of the APOE genotype on brain morphology, function and metabolism, related to other factors such as cognitive reserve, cognition and episodic memory, in subjects at greater risk of developing AD.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the influence of age and the APOE genotype on brain morphology and function, in 700 cognitively healthy individuals, 45 to 75 years old, recruited from an ongoing longitudinal cognition study exploring memory and executive functions (ClinicalTrials.gov ID: NCT01835717).

All subjects have been APOE genotyped and underwent a clinical and cognitive assessment. Within this study, the subjects will be submitted to an MRI scanning protocol including morphological and resting state acquisitions. An identical follow-up MRI session will be performed in 2 years' time. The analyses will be focused on detecting the effect of the APOE allelic variants on the change rate of the neuroimaging variables as well as its interaction with aging.

ELIGIBILITY:
Inclusion Criteria:

* Participant included in the study ClinicalTrials.gov ID: NCT01835717
* APOE genotype obtained before MRI acquisition
* Be willing to perform an MRI and agree to a 2 years longitudinal follow up
* Sign informed consent

Exclusion Criteria:

* Contraindication to MRI scanning: claustrophobia, pacemaker, history of ocular cerclage, heart valves, aneurysm clips and carrying any metal prosthesis incompatible with MRI.
* Incidental MRI findings that result in the images not being included in the study.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population of this study is 45 to 75 years old at the time of inclusion in the parent study (ClinicalTrials.gov ID: NCT01835717), mostly sons and daughters of AD patients.
Sampling Method: Non-Probability Sample
Enrollment: 575 (Actual)
Dates: Start 2014-04; Primary Completion 2015-07 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Hippocampal atrophy | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Juan D Gispert, PhD, Principal Investigator — Barcelonabeta Brain Research Center, Pasqual Maragall Foundation; José L Molinuevo, MD, PhD, Principal Investigator — IDIBAPS, Hospital Clinic de Barcelona, Barcelonabeta Brain Research Center, Pasqual Maragall Foundation
Locations (1):
- Barcelonabeta Brain Research Center, Barcelona, Spain

REFERENCES:
- [Derived] Ingala S, Mazzai L, Sudre CH, Salvado G, Brugulat-Serrat A, Wottschel V, Falcon C, Operto G, Tijms B, Gispert JD, Molinuevo JL, Barkhof F; ALFA Study. The relation between APOE genotype and cerebral microbleeds in cognitively unimpaired middle- and old-aged individuals. Neurobiol Aging. 2020 Nov;95:104-114. doi: 10.1016/j.neurobiolaging.2020.06.015. Epub 2020 Jun 29. PMID 32791423
- [Derived] Brugulat-Serrat A, Rojas S, Bargallo N, Conesa G, Minguillon C, Fauria K, Gramunt N, Molinuevo JL, Gispert JD. Incidental findings on brain MRI of cognitively normal first-degree descendants of patients with Alzheimer's disease: a cross-sectional analysis from the ALFA (Alzheimer and Families) project. BMJ Open. 2017 Mar 24;7(3):e013215. doi: 10.1136/bmjopen-2016-013215. PMID 28341686
- See also: Main home page — https://fpmaragall.org/en/